CLINICAL TRIAL: NCT06437938
Title: The Effects of Dietary Supplements on Glycemic Control, Body Composition and Hepatic Fat Content in People With Prediabetes: a Randomized, Double-blind, Placebo-controlled Pilot Study
Brief Title: The Effects of Dietary Supplements on Glycemic Control, Body Composition and Hepatic Fat Content in People With Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: BIOGENA GmbH (Unknown)
Responsible Party: Principal Investigator, Michael Leutner, Priv.Doz. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1543/2023
Record Dates: First submitted 2024-05-16; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: PreDiabetes
Keywords: Prediabetes; Dietary supplements
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo group 1 (Placebo Comparator): Corresponding to dietary supplement groups B and C
  Interventions: Other: Placebo group 1: Placebo capsules corresponding to DiaPhyt® Formula 3.0/Berberin Phytoactive Gold
- Placebo group 2 (Placebo Comparator): Corresponding to dietary supplement A
  Interventions: Other: Placebo group 2: Placebo powder corresponding to Wasabi leaf powder
- Dietary supplement group A (Experimental): Wasabi leaf powder
  Interventions: Dietary Supplement: Dietary supplement A: Wasabi leaf powder (product of BIOGENA GmbH & Co KG)
- Dietary supplement group B (Placebo Comparator): Berberin Phytoactive Gold
  Interventions: Dietary Supplement: Dietary supplement B: Berberin Phytoactive Gold (product of BIOGENA GmbH & Co KG)
- Dietary supplement group C (Placebo Comparator): DiaPhyt® Formula 3.0
  Interventions: Dietary Supplement: Dietary supplement C: DiaPhyt® Formula 3.0 (product of BIOGENA GmbH & Co KG)

INTERVENTIONS:
Dietary Supplement: Dietary supplement A: Wasabi leaf powder (product of BIOGENA GmbH & Co KG) — To be taken according to the information in the study protocol/patient information leaflet.
  Arms: Dietary supplement group A
Dietary Supplement: Dietary supplement B: Berberin Phytoactive Gold (product of BIOGENA GmbH & Co KG) — To be taken according to the information in the study protocol/patient information leaflet.
  Arms: Dietary supplement group B
Dietary Supplement: Dietary supplement C: DiaPhyt® Formula 3.0 (product of BIOGENA GmbH & Co KG) — To be taken according to the information in the study protocol/patient information leaflet.
  Arms: Dietary supplement group C
Other: Placebo group 1: Placebo capsules corresponding to DiaPhyt® Formula 3.0/Berberin Phytoactive Gold — To be taken according to the information in the study protocol/patient information leaflet.
  Arms: Placebo group 1
Other: Placebo group 2: Placebo powder corresponding to Wasabi leaf powder — To be taken according to the information in the study protocol/patient information leaflet.
  Arms: Placebo group 2

SUMMARY:
This clinical study aims to explore the effects of 3 dietary supplements on metabolic parameters, liver fat content, and body composition in individuals with prediabetes. Prediabetes refers to a condition where blood sugar levels are higher than normal but not high enough for a diabetes diagnosis. The study will last for three months, during which participants will either take a dietary supplement or a placebo. Five groups will be studied, including placebo groups. Blood tests will assess glucose and lipid metabolism parameters, adipokines, and liver and kidney function. Liver stiffness and fat content will also be measured using elastography. Additionally, body composition will be assessed, and participants' psychological state, quality of life, eating habits and sports habits will be evaluated using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* willingness and ability to provide written informed consent and comply with all study requirements,
* age between 40 and 80 years
* prediabetes with a HbA1c level between 5,7-6,4%
* no antidiabetic treatment prior to the inclusion in the study
* BMI between 25 and 35 kg/m2
* fasting glucose of 100-125mg/dl
* in the case of women of childbearing potential, providing a negative pregnancy test at inclusion and once a month until the end of the study

Exclusion Criteria:

* failure to provide written informed consent and/or failure to comply with the study requirements
* age <40 years
* HbA1c outside of the set range
* significant impairments of hepatic and/or renal function
* clinically significant abnormalities in medical history, routine laboratory screening, or in physical examination
* allergies against any of the components of the dietary supplements or the placebo
* type 1 diabetes mellitus, latent autoimmune diabetes in adults, maturity-onset diabetes of the young, gestational diabetes
* pregnancy, lactation
* concurrent treatment with any antidiabetic drug
* concurrent treatment with drugs/dietary supplements that have proven interactions with dietary supplements included in our study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
changes in the time in range | 2 weeks at baseline before start of the dietary supplement, 2 weeks during the last 2 weeks of the 3 month dietary supplement ingestion phase
  time in range measured with continuous glucose monitoring system

SECONDARY OUTCOMES:
changes in HbA1c values | baseline, after 3 months
  HbA1c (glycated haemoglobin) values
changes in fasting glucose concentration | baseline, after 3 months
  fasting glucose concentration
changes in fasting insulin concentration | baseline, after 3 months
  fasting insulin concentration
changes in fasting c-peptide concentration | baseline, after 3 months
  fasting c-peptide concentration
changes in HOMA-IR | baseline, after 3 months
  HOMA-IR calculated as fasting insulin level (micro-units per milliliter) multiplied by the fasting blood glucose level (milligrams per deciliter), dividing the result by 405
changes in parameters of lipid metabolism | baseline, after 3 months
  HDL, LDL, triglycerides, total cholesterol, apolipoprotein B, chylomicrons
changes in the hepatic fat content | baseline, after 3 months
  hepatic fat content
changes in the hepatic fibrosis amount | baseline, after 3 months
  hepatic fibrosis amount
changes in parameters of hepatic function | baseline, after 3 months
  GGT (gamma-glutamyltransferase), GOT (AST, aspartate transaminase), GPT (ALT, alanine transaminase), alkaline phosphatase
changes in bilirubin concentrations | baseline, after 3 months
  bilirubin
changes in the weight | baseline, after 3 months
  weight
changes in the BMI | baseline, after 3 months
  BMI calculated as weight in kilograms divided by the square of height in meters
changes in the anthropometric parameters | baseline, after 3 months
  fat free mass, fat mass
changes in adipokine levels | baseline, after 3 months
  adiponectin, leptin
changes in depressive, anxiety and stress-related symptoms | baseline, after 3 months
  depressive, anxiety and stress-related symptoms assessed using the Depression-Anxiety-Stress Scale
changes in quality of life | baseline, after 3 months
  quality of life assessed using the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No